CLINICAL TRIAL: NCT01460524
Title: Observational Study on the Use of Hypertonic Saline for the Treatment of Bronchiolitis
Brief Title: Nebulized Hypertonic Saline for Bronchiolitis
Status: Completed | Type: Observational
Sponsor: Hôpital Armand Trousseau (Other)
Collaborators: Hopital Universitaire Robert-Debre (Other); Poissy-Saint Germain Hospital (Other); Versailles Hospital (Other); Hôpital Jean Verdier (Other)
Responsible Party: Principal Investigator, CARBAJAL, Professor of Pediatrics, Hôpital Armand Trousseau
Other Study IDs: Bronchiolitis-saline
Record Dates: First submitted 2011-10-25; First posted 2011-10-27 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Bronchiolitis
Keywords: bronchiolitis; saline; nebulization; hypertonic
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In randomized controlled trials, the use of nebulized hypertonic saline in acute bronchiolitis has been reported to improve respiratory distress scores, to reduce length of hospital stay and to show a trend towards lower hospitalization rates.

The investigators aim to verify by an observational study if the rate of hospital admission and the length of hospital stay of infants presenting to the emergency department (ED) with bronchiolitis decreases after the inclusion of 5.85% nebulized hypertonic saline in the treatment strategy of the ED and hospitalization wards.

The investigators will assess the evolution of hospital admission rates and the length of hospital stay in two hospitals that use 5.85% nebulized hypertonic saline for the treatment of bronchiolitis and in two hospital that do not use these nebulizations. If nebulized hypertonic saline is effective in this setting, then the hospitalization rates and length of stay should be lower during the year of hypertonic saline use compared to two previous years when this therapy was not used. These parameters would not be modified in centers that do not use hypertonic saline.

DETAILED DESCRIPTION:
This is a before-after observational study designed to compare the results in terms of hospitalization rate and length of hospital stay between a period when nebulized hypertonic saline was included in the treatment of bronchiolitis in infants versus the two previous years when this therapy was not used in two hospitals. There will not be any randomization.

Physicians have been instructed on the use of hypertonic saline for moderate and severe bronchiolitis in infants but its totally up to them whether to use this nebulization for each particular patient. Two other hospital where nebulized hypertonic saline has never been used and will not be used during the next bronchiolitis epidemics will be the control centers.

The study comprises two periods, one prospective starting on November 2011 and ending in March 2012 and one retrospective including the two previous bronchiolitis epidemics, November 2009-March 2012 and November 2010-March 2011.

During the prospective period a standardized assessment of the respiratory status of each infant will be carried out before and after each hypertonic saline nebulization.

ELIGIBILITY:
Inclusion Criteria:

* All infants up to 1 year of age presenting to the ED for bronchiolitis during the study periods.

Exclusion Criteria:

* Bronchiolitis in infants older than 1 year

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: For the prospective part of the study, all infants up to 1 year of age presenting to the ED for bronchiolitis from November 1st, 2011 to March 30th, 2012 will be included in this observational study. For the retrospective part of the study, data of all infants up to 1 year of age who were seen in the ED for bronchiolitis from November 1st, 2009 and March 30th, 2010 and from November 1st, 2010 and March 30th, 2011 will be analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 2580 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Hospitalization rate | 6 MONTHS
  Comparison of hospitalization rates of infants presenting to the ED with bronchiolitis during the year of use of nebulized hypertonic saline versus the two previous years when nebulized hypertonic saline was not used.

SECONDARY OUTCOMES:
Length of hospital stay | 6 months
  Comparison of lenghts of stay of infants hospitalized for bronchiolitis during the year of use of nebulized hypertonic saline in hospitalization wards versus the two previous years when nebulized hypertonic saline was not used.
Assessment of 5.85% hypertonic saline tolerance | 6 months
  A standardized assessment of the respiratory status will be carried out right before and after each nebulization

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Carbajal, MD, PhD, Principal Investigator — Hôpital Armand Trousseau, Paris
Locations (5):
- France (5):
  - Hôpital de Versailles, Le Chesnay
  - Hôpital Armand Trousseau, Paris
  - Hôpital Robert Debré, Paris
  - CHI Poissy Saint Germain en Laye, Poissy
  - Hôpital Jean Verdier, Bondy, Île-de-France Region